CLINICAL TRIAL: NCT07245472
Title: Clinical Effect of Kinesio Taping Combined With Dry Needling to Myofascial Trigger Point on Shoulder-hand Syndrome in Hemiplegia Patients
Brief Title: The Treatment of Shoulder-hand Syndrome in Hemiplegia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Handan Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HandanCentral
Record Dates: First submitted 2025-09-12; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-09

CONDITIONS: Shoulder-hand Syndrome
Keywords: Shoulder-hand syndrome; Dry Needling; Kinesio Taping; Myofascial Trigger Points
MeSH Terms: conditions — Reflex Sympathetic Dystrophy | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (n = 28) received DN and sham Kinesio taping (Experimental): An experienced physician performed the DN treatment. Active myofascial trigger points (MTrPs) were identified via physical examination in the deltoid, subscapularis, supraspinatus, and infraspinatus muscles. After disinfecting with alcohol, the most painful points were punctured using a sterile 0.3mm × 50mm needle (Hua Tuo, Suzhou Medical Supplies Factory Co., Ltd., China) until a local twitch response (LTR) was elicited. Upon needle removal, the investigators applied pressure with a cotton swab to prevent hematoma. The supraspinatus was needled with the participant seated, while the other muscles were treated in the prone position. For sham taping, the same type of white sports tape as used in Group B was applied-without tension-to the same anatomical area, with the participant's vision blocked.
  Interventions: Device: Dry Needling; Device: Sham Kinesio taping
- Group B (n = 28) was treated with KT and sham DN (Experimental): Participants underwent eight KT applications, each retained for two days, with a two-day interval after every two applications. Standard 5-cm white KT tape was used. The protocol included: an X-shaped strip anchored at the coracoid process with 50-75% tension; an I-shaped strip applied along the supraspinatus muscle with the shoulder extended, adducted, and internally rotated, plus contralateral cervical bending; and two additional I-shaped strips reinforcing the anterior and posterior deltoid using a strengthening technique, with anchors at the outer third of the clavicle and scapula. All tapes ended without tension. The same physician performed all taping. For sham DN, a sterile 0.3×50 mm needle was used at the same MTrP locations as in the DN group, with participants' vision blocked. The sham procedure aimed to produce a tingling sensation without eliciting a local twitch response to maintain blinding.
  Interventions: Device: Kinesio Taping; Device: Sham Dry Needling
- Group C (n = 28) was treated with KT combined with DN. (Experimental): Participants received both active DN and KT interventions
  Interventions: Device: Dry Needling; Device: Kinesio Taping

INTERVENTIONS:
Device: Dry Needling — The deltoid, subscapularis, supraspinatus,and infraspinatus muscles were examined through physical examination to determine the active myofascial trigger points (MTrPs). After disinfection with alcohol, a sterile needle with a diameter of 0.3mm*50mm (China, Suzhou Medical Supplies Factory Co., Ltd.Hua Tuo) was used to puncture the most painful points until a local twitch response (LTR) was obtained. After removing the needle,we pressed it with a cotton swab to prevent local hematoma. The prone position was adopted for the infraspinatus, deltoid and subscapular muscles, and sitting position was adopted for DN treatment of the supraspinatus.
  Arms: Group A (n = 28) received DN and sham Kinesio taping; Group C (n = 28) was treated with KT combined with DN.
Device: Sham Kinesio taping — For the treatment with the sham Kinesio taping, Researchers used the sports white tape of the same specification as the Kinesio taping , and blocked the vision of the participants to apply the same dose as that in Kinesio taping to the same area where the Kinesio taping was applied, so that it could be applied to the skin of the same area where the Kinesio taping was applied without pulling force.
  Arms: Group A (n = 28) received DN and sham Kinesio taping
Device: Kinesio Taping — Patients received eight therapeutic kinesiology taping (KT) sessions. Each application remained for two days, with a two-day interval after every two treatments. Standard 5-cm white KT was used.A 10-cm X-shaped tape was first applied with its center anchored at 50-75% tension over the coracoid process under downward pressure; the tails were laid without tension.A second I-shaped tape was applied with the strengthening technique along the supraspinatus muscle from origin to insertion, with the shoulder extended, adducted, and internally rotated, and the neck contralaterally flexed. The ends (2.5-5 cm) were fixed without tension.The third and fourth I-shaped tapes targeted the anterior and posterior deltoid. With the patient seated, anchors were placed on the lateral clavicle and scapula. The tape was stretched over the deltoid with the shoulder horizontally extended and externally rotated into abduction.
  Arms: Group B (n = 28) was treated with KT and sham DN; Group C (n = 28) was treated with KT combined with DN.
Device: Sham Dry Needling — For sham DN treatment, Researchers used a 0.3mm*50 mm sterile needle (China, Suzhou Medical Supplies Factory Co., Ltd., Hua Tuo) and blocked the participants eyesight with the DN group of the same dose used in the local MTrP of the same area. The effectiveness of the blinding strategy was verified through experiments based on the criterion of causing a tingling sensation without causing LTR.
  Arms: Group B (n = 28) was treated with KT and sham DN

SUMMARY:
The purpose of this clinical study is to investigate effects of Kinesio taping (KT) combined with dry needling (DN) on myofascial trigger points (MTrPs) in post-stroke hemiplegic shoulder-hand syndrome (SHS).

Methods: A prospective, double-blind randomized controlled trial was conducted on 84 SHS patients, who were randomized into three groups: DN (Group A), KT (Group B), and DN+KT (Group C), all receiving standard rehabilitation. VAS, ADL, FMA-UE, PROM, and 8-figure dimensional difference were assessed pre- and post-28-day treatment. Statistical analysis was performed using SPSS 27.0, with paired t-test for intragroup comparisons and independent sample t-test for intergroup comparisons, and statistical significance was set at P<0.05.

DETAILED DESCRIPTION:
A total of 87 patients with stage I shoulder-hand syndrome (SHS) were enrolled between November 2023 and October 2024. Diagnostic criteria followed the Chinese guidelines for acute ischemic stroke (2023) and stroke rehabilitation therapy (2011). Key diagnostic features included unilateral shoulder and hand pain, local skin flushing, increased skin temperature, limited finger flexion, and exclusion of other causes such as trauma or infection. Three participants withdrew, leaving 84 who completed the study.

Participants were randomly assigned to one of three groups (DN, KT, DN+KT) in a 1:1: ratio via a computer-generated random number table (SPSS 27.0). The sequence was concealed using sequentially numbered, sealed opaque envelopes. Group assignment was revealed only to the treating therapist at the time of intervention. Participants and outcome assessors remained blinded throughout the study.

All groups received standard rehabilitation including passive and active range-of-motion exercises, strengthening, and functional training. No analgesics or anti-inflammatory drugs were permitted.

Treatment Group A (n = 28) received DN and sham Kinesio taping: Received dry needling targeting active myofascial trigger points in shoulder muscles, performed by an experienced physician. Sham KT was applied without tension using the same tape as in the KT group.

Group B (n = 28) was treated with KT and sham DN: Received therapeutic Kinesio taping applied in multiple strips with specific tension techniques. Sham DN was performed using a needle without eliciting a local twitch response.

Group C (n = 28) was treated with KT combined with DN: Received both active DN and KT interventions.

ELIGIBILITY:
Inclusion Criteria:

* Within the recovery period from stroke with stable vital signs
* Diagnosis of Stage I shoulder-hand syndrome (SHS)
* SHS onset within 3 months prior to enrollment
* Aged between 40 and 80 years
* Willingness to participate in the trial and provision of signed informed consent

Exclusion Criteria:

* SHS caused by brain trauma or other non-stroke etiologies
* History of shoulder or neck pain due to cervical spondylosis or scapulohumeral periarthritis
* Diagnosis of malignant tumors
* Presence of psychotic disorders or other severe systemic diseases
* Coagulation disorders
* Skin allergies or leukemia contraindicating acupuncture treatment
* Known skin allergy to Kinesio tape
* Concurrent participation in other traditional Chinese medicine or interventional therapies during the trial period
* Joint pain or dyskinesia resulting from peripheral neuropathy

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | Baseline, 14 days, and 28 days post-treatment.
  Pain intensity was assessed using the Visual Analog Scale (VAS). The scale consists of a 10-cm horizontal line with endpoints labeled "0" (no pain) and "10" (worst pain possible). Patients marked their perceived pain level on the line, with scores rounded to the nearest 0.25. Higher scores indicate more severe pain.
Upper Limb Motor Function | Baseline, 14 days, and 28 days post-treatment.
  The simplified Fugl-Meyer Assessment for Upper Extremity (FMA-UE) was used to evaluate upper limb motor function. The total score is 66 points, with higher scores indicating better upper limb motor function.

SECONDARY OUTCOMES:
Degree of Finger Edema | Baseline, 14 days, and 28 days post-treatment.
  Finger swelling was evaluated by measuring the difference in the "8-figure" circumference between the affected and healthy hands. The measurement started from the ulnar styloid process, parallel to the wrist crease, passed around the dorsum of the hand across the fifth and second metacarpophalangeal joints, diagonally crossed the back of the hand, and returned to the starting point.
Passive Range of Motion of the Shoulder Joint | Baseline, 14 days, and 28 days post-treatment.
  Passive range of motion of the shoulder joint was measured using a standard goniometer. Assessment indicators included passive flexion, extension, abduction, adduction, horizontal abduction, horizontal adduction, horizontal medial rotation, and horizontal lateral rotation .
Activities of Daily Living | Baseline, 14 days, and 28 days post-treatment.
  The Activities of Daily Living scale was used for assessment. This scale includes 10 aspects: eating, personal hygiene, bathing, toileting, dressing, anal control, bladder control, bed-chair transfer, level walking, and stair climbing, with a total score of 100 points . A score >60 indicates that the patient can independently perform activities of daily living, with higher scores indicating better living ability.

CONTACTS AND LOCATIONS:
Locations (1):
- Handan Central Hospital, Handan, Hebei, China